CLINICAL TRIAL: NCT06067867
Title: Kidney and Pregnancy Registry
Status: Recruiting | Type: Observational
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Tatiana Besse-Hammer, Head of clinical research unit, Brugmann University Hospital
Other Study IDs: CHUB-BrugKidPreg Reg
Record Dates: First submitted 2023-09-28; First posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-09

CONDITIONS: Kidney Diseases
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Kidney and Pregnancy clinic consultations: Patients followed at the Kidney and Pregnancy clinic pre-conception, during pregnancy and postpartum and patients subsequently referred to nephrological follow-up
  Interventions: Other: Data extraction from medical files

INTERVENTIONS:
Other: Data extraction from medical files — Data extraction from medical files

SUMMARY:
Maternal physiological adaptation to pregnancy plays an important role in the smooth progress of the pregnancy and the healthy growth of the fetus. This physiological adaptation takes place at the level of several organs, including the kidney. Physiological changes during a normal pregnancy take place at the anatomical, glomerular and tubular level.

In the event of pre-existing kidney damage (glomerular and tubular diseases, stone disease, high blood pressure (hypertension) etc...) these adaptations will not be optimal. This will have implications for:

* the course of the pregnancy with the occurrence of feto-maternal complications: miscarriages, pre-eclampsia, intrauterine growth retardation (IUGR), low birth weight, prematurity. The risk of feto-maternal complications increases with the degree of renal failure or with certain pathologies such as lupus.
* progression of kidney disease

Some maternal complications have long-term implications: preeclampsia is associated with a high risk of subsequent cardiovascular and renal complications. Pregnancies in these patients are high-risk pregnancies and require specialized management by an experienced group of gynecologists and nephrologists.

The creation of a retrospective and prospective register by collecting demographic, clinical, biological, radiological and genetic data concerning patients at each consultation within the CHU Brugmann Hospital will allow:

* to establish the epidemiological and clinico-biological characteristics of the patients followed at the Kidney and Pregnancy Clinic at the CHU Brugmann Hospital
* to analyze the risk factors for feto-maternal complications
* to analyze the risk factors for the occurrence of subsequent cardio-renal pathologies in patients who have had preeclampsia or an event during their pregnancy
* to identify patients who will need specialized genetic testing

ELIGIBILITY:
Inclusion Criteria:

1. Pre-conception consultations

   Woman of childbearing age with:
   * Renal damage (glomerular, tubular disease, renal lithiasis, systemic disease, metabolic diseases, congenital diseases, etc.)
   * Hematological disorders (sickle cell disease)
   * Kidney transplantation
   * High blood pressure (hypertension)
   * Pre-kidney transplant assessment in progress for discussion of contraception and pregnancy after kidney transplantation
   * Preeclampsia
   * Multiple miscarriages
   * IUGR and low birth weight in the fetus
   * Family history of kidney disease
2. Peri-gravid consultations

   Pregnant women with
   * Pre-existing kidney damage
   * De novo renal failure (IR)
   * Proteinuria
   * Hematuria
   * Chronic hypertension
   * Pregnancy hypertension
   * Renal lithiasis
3. Postpartum consultations

Postpartum women with

* Early/late pre-eclampsia
* Eclampsia / Hemolysis Elevated Liver enzymes Low Platelet (HELLP) syndrome
* Pregnancy hypertension
* Postpartum hemorrhage
* De novo renal failure postpartum

Exclusion Criteria:

Male patients Menopausal patients

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Patients followed at the Kidney and Pregnancy clinic pre-conception, during pregnancy and postpartum and patients subsequently referred to nephrological follow-up
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-09-12 (Actual); Primary Completion 2043-12 (Estimated); Study Completion 2043-12 (Estimated)

PRIMARY OUTCOMES:
Epidemiological characteristics of patients | 20 years
Clinico-biological characteristics of patients | 20 years
Risk factors for feto-maternal complications | 20 years
Risk factors for cardio-renal pathologies | 20 years
  Risk factors for the occurrence of subsequent cardio-renal pathologies in patients who had preeclampsia or an event during their pregnancy
Need for genetic testing | 20 years
  Identification of patients who will need specialized genetic testing

CONTACTS AND LOCATIONS:
Overall Officials: Christelle Fosso, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No